CLINICAL TRIAL: NCT02257489
Title: A Phase 1, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Local Muscle Injections of ACE-083 in Healthy Postmenopausal Women
Brief Title: Phase 1 Study of ACE-083 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A083-01
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 50 mg single dose (Experimental): 8 subjects in total; 6 subjects to received ACE-083 (50 mg) and 2 subjects to receive placebo, single injection, intramuscularly
  Interventions: Drug: ACE-083
- 100 mg single dose (Experimental): 8 subjects in total; 6 subjects to received ACE-083 (100 mg) and 2 subjects to receive placebo, single injection, intramuscularly
  Interventions: Drug: ACE-083
- 200 mg single dose (Experimental): 8 subjects in total; 6 subjects to received ACE-083 (200 mg) and 2 subjects to receive placebo, single injection, intramuscularly
  Interventions: Drug: ACE-083
- 100 mg multiple dose (Experimental): 8 subjects in total; 6 subjects to received ACE-083 (100 mg) and 2 subjects to receive placebo, two injections 3 weeks apart, intramuscularly
  Interventions: Drug: ACE-083
- 200 mg multiple dose (Experimental): 8 subjects in total; 6 subjects to received ACE-083 (200 mg) and 2 subjects to receive placebo, two injections 3 weeks apart, intramuscularly
  Interventions: Drug: ACE-083
- 100 mg (multiple dose) (Experimental): 9 subjects in total; 6 subjects to received ACE-083 (100 mg) and 3 subjects to receive placebo, two injections 3 weeks apart, intramuscularly
  Interventions: Drug: ACE-083
- 150 mg multiple dose (Experimental): 9 subjects in total; 6 subjects to received ACE-083 (150 mg) and 3 subjects to receive placebo, two injections 3 weeks apart, intramuscularly
  Interventions: Drug: ACE-083

INTERVENTIONS:
Drug: ACE-083 — recombinant fusion protein

SUMMARY:
This study will evaluate the safety and tolerability of single and multiple doses of ACE-083 as a local injection into selected skeletal muscles of healthy subjects. The study will also determine the amount of ACE-083 that reaches the systemic circulation following local administration. Additionally, the study will assess whether local administration into skeletal muscle results in an increase in the size and/or strength of the injected muscle.

DETAILED DESCRIPTION:
ACE-083 is a molecule that has been shown to increase skeletal muscle mass in animals and, therefore, has potential utility in certain diseases that affect skeletal muscle. This initial study in healthy human subjects will help determine the properties of ACE-083 (safety, tolerability, drug absorption and biologic activity), following local administration into skeletal muscle, in advance of clinical trials in patients.

The study will consist of up to 7 planned groups of 8 or 9 subjects each. Subjects in each cohort will be randomized to receive either ACE-083 or placebo. ACE-083 (or placebo) will be administered locally into the right quadriceps (thigh) muscle or right tibialis anterior (lower leg) muscle. Subjects will receive a total of either one dose (on Day 1) or two doses (on Day 1 and Day 22). Each dose administered could include up to 4 injections of study drug into pre-defined locations in the muscle.

A Safety Review Team (SRT) will review blinded, preliminary data from each treatment group to make recommendations regarding escalation to the next treatment group. Subjects will be assessed for safety throughout the treatment and follow-up periods. Follow-up visits will occur over 12 weeks following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, defined by follicle stimulating hormone (FSH) level > 40 IU/L and either 12 months of spontaneous amenorrhea or at least 6 months post-surgical bilateral oophorectomy and/or hysterectomy
* BMI 18.5-32 kg/m2
* Clinical laboratory values that meet the following criteria prior to dosing on Study Day 1: (i) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2 x upper limit of normal (ULN), (ii) Calculated creatinine clearance ≥ 60 mL/min, (iii) Platelet count ≥ 100 x109/L
* Able to adhere to the study visit schedule, understand and comply with protocol requirements
* Understand and sign written informed consent

Exclusion Criteria:

* History of hepatitis B (HBsAg and HB core Ab), human immunodeficiency virus (HIV) antibody or active hepatitis C
* Positive drug or alcohol screen test at screening or on Day 1
* History of drug or alcohol abuse (as defined by the Investigator) or required treatment for drug or alcohol use within 2 years of Day 1
* Donation or loss ≥ 500 mL of whole blood within 2 months prior to Day 1
* History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia) within 6 months prior to screening; serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening
* History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins
* History of active malignancy, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
* History of clinically significant (as determined by the Investigator) cardiac, endocrine, hematologic, hepatic, immune, metabolic, urologic, pulmonary, neurologic, neuromuscular, dermatologic, psychiatric, renal, and/or other disease
* Treatment with systemic glucocorticoid therapy, statin medication, insulin, oral hormone replacement therapy or any other therapy (including investigational) with known or intended effects on muscle within 3 months prior to Day 1
* Treatment with anti-platelet, anti-coagulant, or any other therapy (including investigational) with known or intended effects on bleeding risk within 1 week prior to Day 1
* Treatment with another investigational drug, or approved therapy for investigational use within 4 weeks prior to Day 1, or if the half-life of the previous product is known, within 5 times the half-life prior to Day 1, whichever is longer
* Treatment within 3 months prior to Day 1 with any potent cytochrome P450 (CYP) 3A4/5 inhibitors (e.g., verapamil, ketoconazole, micronazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, delavirdine) or CYP3A4/5 inducers (carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, St. John's wort)
* Subject is unwilling or unable to maintain physical activity at baseline level for the duration of the study
* Subject has any condition that would prevent MRI scanning (e.g., pacemaker, knee/hip replacement, metallic implant, or extreme claustrophobia)
* Subject is unsuitable for enrollment in the opinion of the Investigator or Sponsor for other unspecified reasons

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Manager, Study Director — Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA
Locations (1):
- Acceleron Investigative Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glasser CE, Gartner MR, Wilson D, Miller B, Sherman ML, Attie KM. Locally acting ACE-083 increases muscle volume in healthy volunteers. Muscle Nerve. 2018 Jun;57(6):921-926. doi: 10.1002/mus.26113. Epub 2018 Mar 15. PMID 29486514

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg Single Dose (RF): 8 subjects in total; 6 subjects to receive ACE-083 (50 mg) and 2 subjects to receive placebo, single injection, intramuscularly in the rectus femoris (RF)
  ACE-083: recombinant fusion protein
- 100 mg Single Dose (RF): 8 subjects in total; 6 subjects to receive ACE-083 (100 mg) and 2 subjects to receive placebo, single injection, intramuscularly in the rectus femoris (RF)
  ACE-083: recombinant fusion protein
- 200 mg Single Dose (RF): 8 subjects in total; 6 subjects to receive ACE-083 (200 mg) and 2 subjects to receive placebo, single injection, intramuscularly in the rectus femoris (RF)
  ACE-083: recombinant fusion protein
- 100 mg Multiple Dose (RF): 8 subjects in total; 6 subjects to receive ACE-083 (100 mg) and 2 subjects to receive placebo, two injections 3 weeks apart, intramuscularly in the rectus femoris (RF)
  ACE-083: recombinant fusion protein
- 200 mg Multiple Dose (RF): 8 subjects in total; 6 subjects to receive ACE-083 (200 mg) and 2 subjects to receive placebo, two injections 3 weeks apart, intramuscularly in the rectus femoris (RF)
  ACE-083: recombinant fusion protein
- 100 mg Multiple Dose (TA): 9 subjects in total; 6 subjects to receive ACE-083 (100 mg) and 3 subjects to receive placebo, two injections 3 weeks apart, intramuscularly in the tibialis anterior (TA)
  ACE-083: recombinant fusion protein
- 150 mg Multiple Dose (TA): 9 subjects in total; 6 subjects to receive ACE-083 (150 mg) and 3 subjects to receive placebo, two injections 3 weeks apart, intramuscularly in the tibialis anterior (TA)
  ACE-083: recombinant fusion protein
- Pooled Placebo (RF): Pooled placebo from the rectus femoris (RF) cohorts, n=10 (n=2 from each RF cohort)
- Pooled Placebo (TA): Pooled placebo from the tibialis anterior cohorts, n=6 (n=3 from each TA cohort)
Period: Overall Study
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA) | Pooled Placebo (RF) | Pooled Placebo (TA)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6
Completed | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 10 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA) | Pooled Placebo (RF) | Pooled Placebo (TA) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (4.29) | 54.2 (9.99) | 55.0 (2.37) | 55.2 (3.71) | 57.0 (2.45) | 55.7 (3.08) | 57.0 (4.73) | 59.2 (5.53) | 56.7 (7.50) | 56.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 58
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 5 | 6 | 5 | 6 | 5 | 6 | 10 | 6 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  White | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 10 | 5 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: ACE-083 Safety and Tolerability: Number of Subjects With Adverse Events
Description: Safety/tolerability assessment, following intramuscular administration, includes adverse events, injection site reactions, laboratory measurements, vital signs, etc.
Time Frame: From initiation of treatment (Study Day 1) to end of follow up period (up to Study Day 106)
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA) | Pooled Placebo (RF) | Pooled Placebo (TA)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6
Participants | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6

2. Secondary Outcome: ACE-083 Pharmacokinetics: Maximum Measured Plasma Concentrations
Description: Assessment of systemic absorption and exposure following local injection of ACE-083 into the thigh or lower leg muscle
Time Frame: PK samples were collected predose, and at 3 hours and 6 hours postdose.
Measure: Number; unit: ng/mL (Cmax)
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
ng/mL (Cmax)
  Cmax (min) dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cmax (max) dose 1 | 0 | 168 | 226 | 112 | 219 | 132 | 136

3. Secondary Outcome: ACE-083 Pharmacodynamics
Description: Pharmacodynamic assessments include measurements of thigh or lower leg volume and composition (by MRI) and muscle strength testing (by hand-held dynamometer and fixed system)
Time Frame: From initiation of treatment (Study Day 1) to end of follow up period (up to Study Day 106)
Reporting Status: Not Posted

4. Secondary Outcome: ACE-083 Pharmacokinetics: Time of the Maximum Measured Plasma Concentration
Description: Assessment of systemic absorption and exposure following local injection of ACE-083 into the thigh or lower leg muscle
Time Frame: PK samples were collected predose, and at 3 hours and 6 hours postdose.
Measure: Number; unit: h (Tmax)
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
h (Tmax)
  Tmax (min) dose 1 | 0 | 96 | 96 | 96 | 600 | 24.00 | 96.0
  Tmax (max) dose 1 | 0 | 96 | 168 | 96 | 600 | 96.0 | 96.0

ADVERSE EVENTS:
Arm/Group | 50 mg Single Dose (RF) | 100 mg Single Dose (RF) | 200 mg Single Dose (RF) | 100 mg Multiple Dose (RF) | 200 mg Multiple Dose (RF) | 100 mg Multiple Dose (TA) | 150 mg Multiple Dose (TA) | Pooled Placebo (RF) | Pooled Placebo (TA)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 10/10 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Single Dose (RF) (N=6) | 100 mg Single Dose (RF) (N=6) | 200 mg Single Dose (RF) (N=6) | 100 mg Multiple Dose (RF) (N=6) | 200 mg Multiple Dose (RF) (N=6) | 100 mg Multiple Dose (TA) (N=6) | 150 mg Multiple Dose (TA) (N=6) | Pooled Placebo (RF) (N=10) | Pooled Placebo (TA) (N=6)
Injection site pain (General disorders) | 5 | 5 | 6 | 5 | 6 | 5 | 6 | 10 | 6
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 0
Injection site discomfort (General disorders) | 0 | 1 | 0 | 3 | 0 | 3 | 1 | 1 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection site hypoaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site paresthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 2 | 0 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 2 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 2 | 6 | 6 | 2 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 4
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 3 | 0 | 4 | 2 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other